CLINICAL TRIAL: NCT03596593
Title: Identifying Microsatellite Instability Status From Circulating Tumor DNA in Chinese Patients With Refractory Advanced Solid Tumors: a Large Molecular Epidemiological Investigation
Brief Title: Identifying MSI Status From ctDNA in Chinese Patients With Refractory Advanced Solid Tumors
Acronym: IMPACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IMPACT-China
Record Dates: First submitted 2018-06-27; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Solid Tumor
Keywords: Solid tumor; China; MSI; ctDNA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): A total of 8-10 mL of blood will be collected from this group of patients and used for blood-MSI testing.
  Interventions: Diagnostic Test: SPANOM (identifying MSI status from ctDNA)

INTERVENTIONS:
Diagnostic Test: SPANOM (identifying MSI status from ctDNA) — SPANOM technique, which has been developed by 3D Medicines Inc. Shanghai, China and made it possible to identify MSI status from blood samples, will be used in patients with refractory advanced solid tumors.

SUMMARY:
This is a molecular epidemiological investigation aiming to identify microsatellite instability status from circulating tumor DNA in Chinese patients with refractory advanced solid tumors.

DETAILED DESCRIPTION:
This study is conducted in Chinese patients with advanced refractory metastatic solid tumors. A total of 8-10 mL of blood will be collected from eligible patients and used for extracting circulating tumor DNA. Blood-MSI status will be tested based on SPANOM technique developed by 3D Medicines Inc. Shanghai, China. Patients are encouraged to provide tissues collected from progressive disease for tissue-MSI testing (not required for inclusion).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age≥18 years old.
2. Confirmed malignant solid tumor by histopathology or cytopathology.
3. Colorectal cancer: progression after second-line therapy. Non-colorectal cancer: progression after first-line therapy.
4. Time duration from the last time of anti-cancer treatment to blood sample collection for MSI testing ≥ two weeks or five times half-life period of anti-cancer drugs
5. Signed the informed consent with name and time.

Exclusion Criteria:

1. Hematological malignancy
2. Patients who received immuotherapies.
3. Patients who received blood transfusion within one month before blood collection.
4. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2018-07-11 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of MSI-H across different cancer types in Chinese patients | Two years

SECONDARY OUTCOMES:
Incidence of Lynch syndrome across different cancer types | Two years
Concordance between blood-MSI and corresponding tissue-MSI status | Two years
  In patients who are able to provide tumor tissue samples, concordance between blood-MSI status by SPANOM technique and tissue-MSI status by polymerase chain reaction (PCR) method will be calculated.
  DNA extracted from each tumor tissue will be amplified by standard PCR using six microsatellite loci: NR-21, BA-26, NR-27, BA-25, NR-24, MONO-27. Tumors are designated MSI-H if more than two loci were instable, MSI-L if one locus is instable, and MSS if all loci are stable.

CONTACTS AND LOCATIONS:
Overall Officials: Shen Lin, Professor, Principal Investigator — Peking University
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhenghang Wang, Hao Qin, Mei Wang, et al. SPANOM: A cost-effective method of detecting MSI in ctDNA. ASCO 2018, abstract e24263.